CLINICAL TRIAL: NCT04225481
Title: Evaluation of Enhanced Therapeutic Effect of Adipose Stromal Vascular Fraction Added With Human Platelet Lysate in Treatment of Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: APolLO
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Assessment of the Trophic and Anti-inflammatory Effect of SVF Added With HPL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SVF from healthy subjects from aesthetic plastic surgery: Subjects undergoing plastic surgery as scheduled by clinic routine to obtain waste adipose tissue
  Interventions: Other: isolation of waste material and culturing with different supplement culture media
- OA patients: Subjects undergoing prosthetic surgery as scheduled by clinic routine to obtain waste synovium and cartilage
  Interventions: Other: isolation of waste material and culturing with different supplement culture media

INTERVENTIONS:
Other: isolation of waste material and culturing with different supplement culture media — isolation of waste material and culturing with different supplement culture media

SUMMARY:
Osteoarthritis (OA) is a highly progressive and debilitating joint disease. Recently, it was demonstrated the existence of an important link between OA inflammation and progression of structural changes. Therapy with intra-articular injection of stromal vascular fraction (SVF) holds great promises and its efficacy could be further augmented with the addition of biological adjuvants. In the present project, we aim at demonstrating that human platelet lysate (HPL) increases the intrinsic beneficial properties of SVF on cartilage regeneration and joint environment. Moreover, we want to verify if SVF-conditioned medium (CM) obtained from SVF primed with HPL yields comparable or superior outcomes than whole SVF.

ELIGIBILITY:
Inclusion Criteria:

OA patients

* Subscription of informed consent
* BMI < 30
* age between 55-75 years included
* Kelgrenn-Lawrence equal or superior to grade III
* presence of synovitis
* patients undergoing knee replacement
* suspension of NSAIDs from one week before the surgical procedure according to the standard clinical practice Healthy subjects from aesthetic plastic surgery
* Subscription of informed consent
* BMI < 30
* age between 18-50 years included
* subjects undergoing liposuction and/or abdominoplasty

Exclusion Criteria:

* HCV, HIV, HBV, TPHA infection
* Pregnancy (auto declaration)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects undergoing aesthetic plastic surgery or OA patients undergoing prosthetic surgery
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Expression of trophic-related genes in cartilage samples treated with SVF added or not with HPL | surgery as scheduled by clinic routine
  With this project, we expect to demonstrate that HPL increases the beneficial properties of SVF on cartilage regeneration and joint environment. We envision that HPL will increase expression of genes involved in ECM synthesis, thus enhancing cartilage regeneration. Based on previous published data, we will consider as statistical a difference between treated (SVF + HPL) and not treated samples (SVF) of two folds in expression of genes involved in ECM production (e.g. COL2A1, ACAN, SOX9). A fold increase equal to 2 is the minimum value to consider biologically relevant the influence of the treatment compared to a control group in which the gene expression is considered to be equal to 1. If our hypothesis will be confirmed, this will allow to improve the current therapy for OA with a biological adjuvant that reduces disease progression and helps cartilage regeneration.

IPD SHARING:
Plan to Share IPD: Undecided